CLINICAL TRIAL: NCT00625755
Title: A Phase I/II Study to Assess the Safety and Efficacy of Vaccinations With Allogeneic Dendritic Cells: Autologous Tumor-Derived Cells Subjected to Electrofusions in Patients With AJCC Stage IV Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, David Avigan, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P001539; DCREN-005-01
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; AJCC Stage IV (primary or relasped) renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Electrofusion DC vaccine — To assess the safety and efficacy of vaccinations

SUMMARY:
This study will look how using taken from your tumors and mixed with special immune stimulating cells from another person's blood in given back to you in a series "fusion cell" injections, will effect your body. The primary goal of the study is to see if giving the experimental fusion cell injections is safe. We will also be looking to see what effect the experimental treatment as on your immune system and whether it has an effect on your cancer.

DETAILED DESCRIPTION:
Patients undergo tumor aquisition and short-term tumor cell cultures are established. Leukopheresis is performed monocyte-derived DC are generated ex-vivo by standard culture techniques, utilizing GM-CSF and Il-4. PEG fusions are generated, and following irradiation, the vaccine is frozen. The thawed vaccine is administered SC into a single site every three weeks. Each study is examining a dose-escalating strategy based apon the number PEG-fused generated from the PEG process that expressed both tumor cell and DC markers as determined by immune staining.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be _> 18 years of age
* The patient must be diagnosed with AJCC stage IV (primary or relasped) RCC
* The patient must have a baseline Eastern Cooperative Oncology Group (ECOG) Clinical performance of 0-1
* The patient must have accessible tumor (minimum of 2.5cm in diameter in aggregate and accessible) for vaccine production
* The patient must have measurable tumor lesions (using Response Evaluation Criteria in Solid Tumors (RECIST) following resection of tumor lesions(s) used for vaccine production. If the patient has received previous radiation or intra-tumoral investigational treatments, the measurable disease must be outside the previous radiation port or treatment area unless there is documented tumor progression following the completion of therapy.
* The patient must have adequate hematologic, hepatic, and renal function parameters within 21 days prior to the first vaccination (day 0 of treatment):

  * White blood cell(WBC) count >_ 3,000 cell/mm3
  * Platelet count >_ 100,000 platelets/mm3
  * Creatine(serum) <2.0mg/dL
  * Total bilirubin <2.0 mg/dL
  * Serum glutamic pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) <2.0 x Upper limits of normal
  * Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) < 2.0 x Upper limits of normal
* The patient must be serologically negative for human immunodeficiency virus (HIV)-1, HIV-2, and human T lymphotropic virus (HTLV)-1
* Female patients of childbearing potential must have negative pregnancy tests, refrain from nursing and must agree ton use appropriate contraception for the duration of the trial
* The patient must have signed and dated written informed consent prior to any study procedures. The consent process must be documented in the patient's medical record

Exclusion Criteria:

* The patient has received prior chemotherapy
* The patient's tumor-derived cells do not meet predetermined manufacturing specifications, for example: human leukocyte antigen (HLA) Class 1 molecule expression, sufficient tumor derived cells for vaccine manufacture, or pathologic confirmation of RCC
* The patient has received more than 2 prior regimes for treatment of RCC and the most recent is within 2 weeks of the first screening procedure
* The patient has received radiation therapy within 2 weeks of the first sceeening procedure
* The patient has a clinically significant autoimmune diorder
* The patient has an active infection at the time of the first screening procedure requiring parenteral antibiotics
* The patient has clinically significant hematolgic, cardiac, renal, or hepatic disease or any other underlying condition that would contraindicate study therapy or confuse interpretation of study results
* The patient has any active or clinically significant central nervous system (CNS) metastases
* The patient has a previous unrelated malignancy or second malignancy within 5 years prior to the first screening procedure, except from non-melanoma skin cancer and in situ carcinomas
* The patient is receiving chronic immunosuppressive, and/or oral steriod treatment
* The patient has any other reason in the Investigator's opinion that would make protocol compliance unmanageable or may compromise the patient's ability to give informed consent
* The patient has been treated with a non-oncologic investigational drug, biologic or medical device within 30 days of the first screening procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-12; Primary Completion 2005-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety of 3 serial vaccinations with allogeneic DCs: autologous tumor-derived cells subjected to electrofusion in patients with AJCC stage IV RCC | screening/baseline, treatment period, follow-up and long-term follow-up

SECONDARY OUTCOMES:
To determine if 3 serial vaccinations of allogeneic DCs: autologous tumor-derived cells subjected to electrofusion will induce a clinical response as assessed by tumor response and will induce an immune response. | screening/baseline, treatment period, follow-up and long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- [Result] Avigan DE, Vasir B, George DJ, Oh WK, Atkins MB, McDermott DF, Kantoff PW, Figlin RA, Vasconcelles MJ, Xu Y, Kufe D, Bukowski RM. Phase I/II study of vaccination with electrofused allogeneic dendritic cells/autologous tumor-derived cells in patients with stage IV renal cell carcinoma. J Immunother. 2007 Oct;30(7):749-61. doi: 10.1097/CJI.0b013e3180de4ce8. PMID 17893567